CLINICAL TRIAL: NCT03375788
Title: Growth Hormone Releasing Hormone Analog to Improve Nonalcoholic Fatty Liver Disease and Associated Cardiovascular Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Takara Stanley, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DK114144 (NIH)
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity; Obesity, Abdominal; Liver Fat; Fatty Liver
Keywords: tesamorelin; obesity; fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Obesity, Abdominal; Fatty Liver | interventions — tesamorelin; Growth Hormone-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled phase for first 12 months, followed by open-label phase for 6 months during which all participants receive active medication (tesamorelin)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tesamorelin (Experimental): tesamorelin (brand name Egrifta) 2mg daily given subcutaneously
  Interventions: Drug: Tesamorelin
- Placebo (Placebo Comparator): identical placebo given subcutaneously daily
  Interventions: Drug: Identical Placebo

INTERVENTIONS:
Drug: Tesamorelin — Tesamorelin F4 formulation 1.4mg daily
  Other Names: Egrifta, TH9507, Growth Hormone Releasing Hormone Analog
  Arms: Tesamorelin
Drug: Identical Placebo — Placebo injection daily
  Arms: Placebo

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is common in individuals with obesity and is a significant threat to public health, because it can lead to impaired liver function and liver failure. Growth hormone is a hormone produced in the pituitary gland that helps regulate metabolism and growth. Individuals with obesity, on average, secrete less growth hormone than individuals without obesity. There are data to suggest that growth hormone may help to reduce the amount of fat in the liver, and may also reduce inflammation in the liver, both of which would be helpful to individuals with NAFLD. The purpose of this study is to investigate whether treatment with a drug called tesamorelin, which is a growth hormone releasing hormone analogue, will decrease liver fat and improve liver inflammation and scarring in obese individuals with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-65yo
2. Body mass index (BMI) ≥ 30kg/m2, or, for participants with known steatohepatitis, BMI ≥ 25kg/m2
3. Hepatic steatosis as demonstrated by either a) Grade 1+ steatosis on a liver biopsy performed within 12 months of the baseline visit, without >10% reduction in body weight or addition of medications to treat fatty liver, or b) liver fat fraction ≥5% on hydrogen-magnetic resonance spectroscopy (1H-MRS)
4. Hepatitis C antibody and Hepatitis B surface antigen negative. Subjects without known history of Hepatitis C or Hepatitis C treatment who have a positive Hepatitis C antibody but a negative hepatitis C viral load will also be eligible.
5. For females ≥50yo, negative mammogram within 1 year of baseline
6. If use of vitamin E ≥400 international units daily, stable dose for ≥6 mos
7. Up to date with colon cancer screening recommended by the participant's primary care physician, using whatever methodology the primary physician recommends. This will be ascertained by self-report. (If a participant does not have a primary care physician, we will discuss that colon cancer screening is recommended, typically starting at age 50y, and refer the participant to primary care through Partners if s/he desires.)

Exclusion Criteria:

1. Heavy alcohol use defined as consumption of > 20 grams daily for women or > 30 grans daily for men for at least 3 consecutive months over the past 5 years assessed using the Lifetime Drinking History Questionnaire
2. Known diagnosis of diabetes, use of any anti-diabetic medications (including thiazolidinediones or metformin), fasting glucose >126mg/dL, or hemoglobin A1c (HbA1c) ≥6.5%. Participants with stable use of metformin ≥6 months will be permitted if it is being used for pre-diabetes or another non-diabetes indication (e.g., PCOS).
3. Use of any specific pharmacological treatments for NAFLD/nonalcoholic steatohepatitis except vitamin E
4. Known cirrhosis, Child-Pugh score ≥7, stage 4 fibrosis on biopsy, or clinical evidence of cirrhosis or portal hypertension on imaging or exam. If a subject is not known to be cirrhotic at screen but is found to be cirrhotic based on the results of liver biopsy at baseline, this subject will be referred to a hepatologist for clinical care and will be excluded from further participation in the study.
5. Chronic systemic corticosteroid use in the ≤6 months prior to the baseline visit
6. Chronic use of Actigall, methotrexate, amiodarone, or tamoxifen
7. Known diagnosis of alpha-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, or autoimmune hepatitis
8. Use of growth hormone or growth hormone releasing hormone within the past 6 months
9. Change in lipid lowering or anti-hypertensive regimen within 2 months of screening
10. Hemoglobin < 10.0 g/dL or Creatinine >1.5mg/dL
11. Active malignancy
12. For men, history of prostate cancer or evidence of prostate malignancy by prostate specific antigen (PSA) > 5 ng/mL
13. Severe chronic illness judged by the investigator to present a contraindication to participation
14. History of hypopituitarism, head irradiation or any other condition known to affect the GH axis
15. Use of physiologic testosterone (men) or estrogen or progesterone (women) unless stable use for a year or more prior to study entry
16. Routine magnetic resonance imaging (MRI) exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clip
17. Weight loss surgery within 1 year before baseline. Weight loss surgery more than 1 year prior to baseline visit is permissible as long as no active weight loss (<10% decrease in weight over past 6 months)
18. For women, positive urine pregnancy test (hCG), trying to achieve pregnancy, or breastfeeding
19. For women able to become pregnant, unwillingness to use an acceptable form of birth control during the study.
20. Known hypersensitivity to tesamorelin or mannitol
21. Contraindication to receiving beta-blocker or nitroglycerin (which are part of the coronary angiography)
22. Significant radiation exposure, including any history of radiation therapy, or any of the following in the 12 months prior to randomization: a) more than 2 percutaneous coronary interventions; b) more than 2 myocardial perfusion studies; 3) more than 2 computed tomography angiograms
23. Active consideration for a procedure or treatment that involves significant radiation exposure as defined above in the 12 months following randomization
24. Not willing or able to adhere to dose schedules and required procedures per protocol
25. Judged by the investigator to be inappropriate for the study for other reasons not detailed above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Final Research Data, with all patient identifiers removed, will be available to other researchers through request to the PI. Because information contained in the final research data will include multiple demographic and biological variables that could potentially be used in concert to identify participants, it will be shared only under a Data Sharing Agreement that includes (1) a commitment to using the data only for research purposes and not to identify any individual participant and (2) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Period: 12-month Double-blind Phase
Arm/Group | Tesamorelin | Placebo
Started | 26 | 25
Completed (Indicates completion of 12 month, double-blind phase and at least one assessment at 12 month visit; primary and key secondary endpoints were measured at the 12 month visit. Please note that the 6-month open-label extension was for longer-term safety rather than efficacy endpoints. Thirty participants continued into these phase, for whom safety data are reported in the adverse effects section.) | 19 | 19
Not Completed | 7 | 6
Period: 6 Month Open Label Phase
Arm/Group | Tesamorelin | Placebo
Started | 17 | 13
Completed | 16 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesamorelin | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10) | 47 (11) | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 15 | 38
  Black | 2 | 1 | 3
  Other | 0 | 7 | 7
  Hispanic ethnicity | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Liver Fat Content
Description: Liver Fat Content as measured by hydrogen-magnetic resonance spectroscopy. All available data used; data not available for 1 participant in tesamorelin group and 3 participants in placebo group.
Time Frame: change from baseline to 12 months
Measure: Median (Inter-Quartile Range); unit: percent change in hepatic fat fraction
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 18 | 16
percent change in hepatic fat fraction | -5.3 [-13.0 to -1.4] | 3.6 [-6.2 to 7.9]

2. Secondary Outcome: NAFLD Activity Score
Description: Nonalcoholic Fatty Liver Disease Activity Score (NAS, scored between 0-8, with higher indicating more severe disease) from liver biopsy. All available data used; data not available for 3 participants in placebo group and 1 participant in tesamorelin group.
Time Frame: change from baseline to 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 0 [-2 to 0] | 0 [-1 to 1]

3. Secondary Outcome: Low Density Lipoprotein (LDL) Cholesterol
Description: All available data utilized. Data not available for 2 participants in tesamorelin group and 3 participants in placebo group.
Time Frame: change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 17 | 16
milligrams per deciliter | -5.7 (27) | -0.7 (16)

4. Secondary Outcome: C-reactive Protein
Description: All available data utilized. Data not available for 2 participants in placebo group.
Time Frame: change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 19 | 17
milligrams per liter (mg/L) | -0.9 (4.2) | 0.0 (4.1)

5. Secondary Outcome: Fibrosis Score
Description: fibrosis score from liver biopsy; all available data used - data not available for 1 participant in tesamorelin group and 3 participants in placebo group. Fibrosis stage scored from 0-4, where 0 indicates no fibrosis and 4 indicates most severe fibrosis, which is cirrhosis.
Time Frame: change from baseline to 12 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tesamorelin | Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 0 [0 to 1] | 0 [0 to 0.5]

ADVERSE EVENTS:
Time Frame: Adverse events for the double-blind phase occurred during months 0-12 of the study (12-month double-blind phase). Adverse events for the open-label phase occurred during months 12-18 of the study (6-month open label phase that occurred at the end of the 12- month double-blind phase).
Groups:
- Double-blind Phase: Tesamorelin: tesamorelin (brand name Egrifta) 2mg daily given subcutaneously for first 12 months
  Tesamorelin: Tesamorelin F4 formulation 1.4mg daily
- Double-blind Phase: Placebo: identical placebo given subcutaneously daily for first 12 months
  Identical Placebo: Placebo injection daily
- Open Label Phase: all patients receiving open-label tesamorelin from months 12-18
Arm/Group | Double-blind Phase: Tesamorelin | Double-blind Phase: Placebo | Open Label Phase
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/26 | 3/25 | 0/30
Other Adverse Events (participants affected / at risk) | 22/26 | 15/25 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Phase: Tesamorelin (N=26) | Double-blind Phase: Placebo (N=25) | Open Label Phase (N=30)
rotator cuff surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | NA
appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | NA
major depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | NA
elective knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | NA
liver hematoma following biopsy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Phase: Tesamorelin (N=26) | Double-blind Phase: Placebo (N=25) | Open Label Phase (N=30)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1) | 2 (3)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Concussion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 6 (9) | 1 (1) | 1 (1)
elevated gamma glutamyl transferase (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Galactorrhea (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointeritis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Injection site bruising (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Injection site erythema (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0) | 3 (3)
Injection site itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site redness (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site stinging (Skin and subcutaneous tissue disorders) | 8 (12) | 1 (3) | 9 (10)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mild loss of coordination (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (unspecified) (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Injection site complaints, other (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 6 (6)
Pain following liver biopsy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebral fractures (from fall) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lower extremity venous thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Wisdom teeth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Interpretation of changes in biopsy data are limited by relatively small sample size as well as the requirement for steatosis but not steatohepatitis at baseline. In other words, not all participants had steatohepatitis or fibrosis at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT03375788/Prot_SAP_000.pdf